CLINICAL TRIAL: NCT06167564
Title: Development of a Diagnostic Test System Based on Microchip Technology for the Detection of IgE-dependent Allergic Reactions
Brief Title: Allergy Diagnostic Test Based on Microchip Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IBCE_Allergytest
Record Dates: First submitted 2023-10-20; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Allergy; Allergy;Food; Allergy Pollen; Allergy Drug
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity; Rhinitis, Allergic, Seasonal; Drug Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Group of adult participants with IgE-dependent allergic reactions. Routine blood serum IgE levels will be compared with the newly developed microarray-based diagnostic test system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine allergy tests (Active Comparator): Routine allergy tests (prick tests, specific IgE detection) will be done to establish the sensibilization of the patient.
  Interventions: Diagnostic Test: Routine allergy tests
- Newly developed microarray-based diagnostic test system (Experimental): Newly developed microarray-based diagnostic test system will be used to establish the sensibilization of the patient.
  Interventions: Diagnostic Test: Newly developed microarray-based diagnostic test system

INTERVENTIONS:
Diagnostic Test: Routine allergy tests — Prick test, specific IgE detection
  Arms: Routine allergy tests
Diagnostic Test: Newly developed microarray-based diagnostic test system — Newly developed microarray-based diagnostic test system for the detection of the specific IgE
  Arms: Newly developed microarray-based diagnostic test system

SUMMARY:
The purpose of this study is to develop a microarray-based diagnostic test system for the determination of allergen specific IgE in human blood serum.

DETAILED DESCRIPTION:
The purpose of this study is to develop a microarray-based diagnostic test system for the determination of allergen specific IgE in human blood serum samples and to assess the sensitivity and specificity of the developed system.

ELIGIBILITY:
Inclusion Criteria:

* Type I allergy (food, drug, pollen)
* The patient can read, understand, follow the examination procedures and complete, if necessary, the required documentation
* Written informed consent

Exclusion Criteria:

* Acute or chronic diseases in the stage of decompensation (except allergy)
* Chronic infectious diseases: HIV, viral hepatitis B, C, tuberculosis
* Patients who are pregnant, breastfeeding
* Chronic and protracted mental disorders, all diseases with the presence of the syndrome of dependence on alcohol, drugs and psychoactive substances, any other condition that makes the patient unable to understand the nature, extent and possible consequences of the study or, in the opinion of the researcher, prevents the patient from observing and performing protocol
* Patients are unable or unwilling to give written informed consent and / or follow research procedures
* Any other medical condition that, in the opinion of the investigator, may be associated with an increased risk to the patient or may affect the outcome or evaluation of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum IgE levels of the specific pollen allergens | 1 month
  Serum IgE levels of the specific pollen allergens will be sudied

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Director — IBCE; Antonina Osipova, Dr, Study Director — IBCE; Ekaterina Shamova, r, Principal Investigator — IBCE
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus